CLINICAL TRIAL: NCT05563402
Title: "Evaluation of Usability and Safety of the Self-balancing Walking System Atalante in Patients With Multiple Sclerosis"
Acronym: EXO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Multiple Sclerosis Center of Catalonia (Other)
Responsible Party: Principal Investigator, Edwin Roger Meza Murillo, Principal Investigator, Multiple Sclerosis Center of Catalonia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PR(AG)285/2022
Record Dates: First submitted 2022-09-19; First posted 2022-10-03 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Multiple Sclerosis; Ataxia; Paraplegia
Keywords: exoskeletons; bioengineering; biomechanics;; biomechatronics;; rehabilitation robotics; Atalante
MeSH Terms: conditions — Multiple Sclerosis; Ataxia; Paraplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): Therefore, the investigators propose an, open, non-randomized study. This study protocol includes 12 one-hour RAGT training sessions for 4 weeks, three times a week, under the supervision of a qualified rehabilitation team.
  Informed consent will be obtained from patients before inclusion in the study, which will be carried out in accordance with the Declaration of Helsinki.
  With the aim of describing Usability as the main objective, and Safety as a secondary objective and functional changes at the level of balance, walking speed and quality of life.
  Interventions: Device: Atalante

INTERVENTIONS:
Device: Atalante — Atalante Gait training: Using the Atalante System (self-reliant walking system), participants will be secured with the appropriate sized harness and attached to an overhead body-weight support system. Each session will begin with a 3-5 minute warm-up in the continuous passive mode (cadence ~40-45 steps/minute).

SUMMARY:
Multiple sclerosis (MS) is the most prevalent chronic inflammatory disease of the central nervous system (CNS), affecting more than 2 million people worldwide,1 it is a degenerative disease that selectively affects the central nervous system and represents the main cause of non-traumatic disability in young adults.

Gait and balance disturbances in MS are common even in the early stages of the disease. Half of the patients report some alteration in the quality of walking within the first month after diagnosis, reaching 90% after 10 years of evolution. 4 5 In addition, it is the symptom to which patients give the most importance 6 and the one that most conditions their activity and participation. 7 The causes of gait disturbance are multifactorial and are influenced by different aspects such as muscle strength, balance, coordination, proprioception, vision, spasticity, fatigue and even cognitive aspects4.

There are multiple interventions, including aerobic, resistance training, yoga, and combined exercise, that have shown significant improvements in walking endurance, regardless of outcome measures (six-minute walking test (6MWT), two-minute walking test 2MWT). 8

In recent years, evidence has been growing around rehabilitation with robotic equipment in people with multiple sclerosis (PwMS), in their study Ye et al. concluded that robotic locomotor training has limited impact on motor functions in multiple sclerosis, but improves fatigue and spasticity, is safe and well-tolerated for PwMS, and less demanding for physical therapists.10 Bowman et al. concluded that robot-assisted gait therapy (RAGT) improves balance and gait outcomes in a clinically significant way in PwMS, RAGT appears more effective compared to non-specific rehabilitation, while showing similar effects compared to non-specific rehabilitation. specific balance and gait training in studies with level 2 evidence. RAGT has several advantages in terms of patient motor assistance, training intensity, safety and the possibility of combining other therapeutic approaches and should be promoted for PwMS with disability in a multimodal rehabilitation setting as an opportunity to maximize recovery.11 In this setting, more larger-scale and better-designed studies with longer training duration and more studies evaluating satisfaction, usability, and effectiveness are needed. of RAGT.

DETAILED DESCRIPTION:
Therefore, the investigators propose an open, non-randomized, pseudo-experimental study.

This study protocol includes 12 one-hour RAGT training sessions for 4 weeks, three times a week, under the supervision of a qualified rehabilitation team.

Informed consent will be obtained from patients before inclusion in the study, which will be carried out in accordance with the Declaration of Helsinki.

With the aim of describing Usability as the main objective, and Safety as a secondary objective and functional changes at the level of balance, walking speed and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, between 18 and 65 years of age
* Confirmed diagnosis of MS
* Expanded Disability Status Scale (EDSS) de Kurtzke from 6.0 to 7.0
* Able to verticalize on a daily basis
* Stable course of disease-modifying therapy over the past 6 months
* Clinical comorbidity asymptomatic (i.e., no underlying cardiovascular disease)
* Height: between approximately 1.60 and 1.90 m.
* Willingness to visit the Multiple Sclerosis Center of Catalonia (CEMCAT) for testing and training.
* Gait disorder conditioned by paresis or hemiparesis associated with ataxia or sensory problems
* Patient having given written consent

Atalante is able to accommodate the following limb lengths:

* Thigh: 380-460mm
* Distance between the ground and the joint space of the knee (to be measured while wearing the shoes they intend to wear with Atalante):

  * 457-607mm for patient with an ankle dorsiflexion ≥ 16°
  * 457-577mm for patient with an ankle dorsiflexion between 13° et 16°
  * 457-567mm for patient with an ankle dorsiflexion between 10° et 13°
  * 457-557mm for patient with an ankle dorsiflexion between 0° and 10°
* Hip with less or equal to 460mm when seated
* Maximum weight:90 kg

Exclusion Criteria:

* Pregnancy
* Starting or switching from fampridine (Fampyra®) in the last 4 weeks
* Height and weight outside the secure standard of safe use, described in the safety guides
* Contraindications to training with Atalante (eg, bone instability, history of osteoporosis or osteoporotic fractures)
* Subjects under Corticosteroids treatment or relapse
* Changes in disease-modifying and symptomatic therapy for MS during the study period
* Subjects with psychiatric or cognitive comorbidities that may interfere with the trial
* Whose joint centers cannot be aligned Atalante's
* Ranges of motion below:

  * Knee: 5° extension, 110° flexion
  * Ankle: 0° dorsiflexion, 9° plantar flexion, 18° inversion and eversion
  * Hip: 115° flexion, 15° extension, 17° abduction, 10° adduction, 10°
  * medial rotation, 20° lateral rotation
* Severe spasticity (greater than Ashworth 3) or uncontrolled clonus
* Severe concurrent medical diseases: infections, circulatory, heart or lung, pressure sores
* Active implantable medical device

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
To describe usability of Robotic-Assisted Gait therapy (RAGT) using the Atalante self-balance exoskeleton for persons with multiple sclerosis (PwMS) and explore patient characteristics related to this feature. | 4 months
  Defining usability as a quality attribute that evaluates the ease of use of user interfaces, evaluating the perspective of patients by the Satisfaction Quebec user Evaluation of Satisfaction with assistive technology (QUEST) score and a questionnaire specific to the use of Atalante device.
  Defining high Usability as: Obtaining a positive score greater than or equal to 70% of the total possible score on the Satisfaction Quebec user Evaluation of Satisfaction with assistive technology (QUEST) score.

SECONDARY OUTCOMES:
To describe safety and occurrence of adverse effect of Robotic-Assisted Gait therapy (RAGT) using the Atalante self-balance exoskeleton for persons with multiple sclerosis (PwMS). | 4 months
  • Defining a low occurrence as the appearance of an adverse effect related to the rehabilitation program in less than 10% of the reported patients. Defining an adverse event later in the chapter on instructions for reporting adverse events
To describe safety of Robotic-Assisted Gait therapy (RAGT) using the Atalante self-balance exoskeleton for persons with multiple sclerosis (PwMS), measured by the occurrence of pressure ulcers | 4 months
  • The occurrence of pressure ulcers more than grade 1 in more than 10% of reported patients. Not taking into account the pressure zones that can be considered as an acceptable effect within the program as long as it is reversible in minutes after the program.
To describe the effect at the functional level of RAGT using the Atalante self-balance exoskeleton for improving Balance outcome. | 4 months
  • Balance: Assess the effect of RAGT at the balance outcome measured by the Berg scale, considering a clinically relevant change for improvement in balance as measured by Berg scale was +3 points, meaning that PwMS are likely to perceive that as a reproducible and clinically important change in them balance performance.21
To describe the effect at the functional level of RAGT using the Atalante self-balance exoskeleton for improving Walking speed, quality of life, depression. | 4 months
  • Walking speed: Assess the effect of RAGT at the walking speed measured by the ten-meters walking test (10-MWT), considering a clinically relevant change as an improvement of 20% of the score with respect to the baseline assess.
To describe the effect at the functional level of RAGT using the Atalante self-balance. Physiological Changes at Bowel Dysfunction | 4 months
  • Physiological Changes: Observe the effect of RAGT at the bowel function using the Neurogenic Bowel Dysfunction Spanish version,
To describe the effect at the self-perception and psychological level of RAGT using the Atalante self-balancing exoskeleton to improve quality of life. | 4 months
  • Using the Multiple Sclerosis Quality of Life-54 Survey Spanish version
To describe the effect at the self-perception and psychological level of RAGT using the Atalante self-balancing exoskeleton to improve quality of life and depression. | 4 months
  • Hospital Anxiety and Depression Scale considering a clinically relevant change of 1.7 points

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Montalban, PHD, Study Director — Multiple Sclerosis Center of Catalonia; Carmen Tur Gomez, PHD, Study Director — Multiple Sclerosis Center of Catalonia
Locations (1):
- Centre d'Esclerosi Mútiple de Catalunya (Cemcat) - Barcelona, Hospital Universitari Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2022-08-10): https://cdn.clinicaltrials.gov/large-docs/02/NCT05563402/Prot_000.pdf